CLINICAL TRIAL: NCT04714528
Title: Physical Activity as Treatment for Depression and Anxiety Towards Affordable Preventive Healthcare - a Randomised Controlled Study (RCT)
Brief Title: Physical Exercise for Treatment of Depression and Anxiety - RCT
Acronym: FYPO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Örebro University, Sweden (Other); Uppsala University (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Yvonne Freund-Levi, Associate Professor, M.D., Ph.D, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 273723
Record Dates: First submitted 2020-11-06; First posted 2021-01-19 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Depression; Anxiety
Keywords: Post Traumatic Stress Disorder; Attention Deficit Hyperactivity Disorder; Exercise; Bipolar disorder; Cognitive functions; Biomarkers; Fatty acids; Cytokines; Neurotrophins; Accelerometer; Microbiota; Metabolomics; Lipidomics
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Attention Deficit Disorder with Hyperactivity; Motor Activity; Bipolar Disorder | interventions — Exercise; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Exercise Group (Active Comparator): 45 minutes of aerobic, high intensity group training, three times per week during a 12-week period.
  Interventions: Other: Physical Exercise
- Relaxation Group (Other): 45 minutes of relaxation therapy once per week for 12 weeks.
  Interventions: Other: Relaxation Therapy

INTERVENTIONS:
Other: Physical Exercise — Physical exercise as described before.
  Arms: Physical Exercise Group
Other: Relaxation Therapy — Relaxation therapy as described before.
  Arms: Relaxation Group

SUMMARY:
In a 12 week randomly controlled open trial 102 participants with symptoms of depression and/or anxiety will be exposed to either aerobic high intensity training (HIT) or relaxation therapy. Cognitive functions, biomarkers, psychiatric symptom scales and physical status will be collected at baseline, after 12 weeks and after a year. Depression and anxiety will be measured twice during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Score ≥12 on MADRS or score ≥16 on BAI
* Inhabitant i Örebro County, Sweden
* BMI ≥18 kg/m^2

Exclusion Criteria:

* Diagnosis of chronic psychotic disease or ongoing psychotic episode.
* Ongoing manic state of bipolar disorder
* Severe somatic disease or condition where high intensity exercise is contraindicated
* Difficulty with reading, hearing or understanding the Swedish language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptom improvement in depression | Change of the score from the baseline to the score at 12 weeks.
  Improvement of symptom severity grade are assessed with Montgomery-Åsberg Depression Rating Scale (MADRS). The minimum and the maximum score is 0 and 60 respectively, and the higher score means a worse outcome.
Symptom improvement in depression | Change of the score from the baseline to the score at 1 year.
  Improvement of symptom severity grade are assessed with Montgomery-Åsberg Depression Rating Scale (MADRS). The minimum and the maximum score is 0 and 60 respectively, and the higher score means a worse outcome.
Symptom improvement in anxiety | Change of the score from the baseline to the score at 12 weeks.
  Improvement of symptom severity grade are assessed with Beck Anxiety Inventory (BAI). The minimum and the maximum score is 0 and 63 respectively, and the higher score means a worse outcome.
Symptom improvement in anxiety | Change of the score from the baseline to the score at 1 year.
  Improvement of symptom severity grade are assessed with Beck Anxiety Inventory (BAI). The minimum and the maximum score is 0 and 63 respectively, and the higher score means a worse outcome.
Subjective symptom improvement in depression | Change of the score from the baseline to the score at 12 weeks.
  Improvement of symptom severity grade are assessed with Montgomery-Åsberg Depression Rating Scale Self-Rating Version (MADRS-S). The minimum and the maximum score is 0 and 60 respectively, and the higher score means a worse outcome.
Subjective symptom improvement in depression | Change of the score from the baseline to the score at 1 year.
  Improvement of symptom severity grade are assessed with Montgomery-Åsberg Depression Rating Scale Self-Rating Version (MADRS-S). The minimum and the maximum score is 0 and 60 respectively, and the higher score means a worse outcome.

SECONDARY OUTCOMES:
Cognitive function: Trail Making Test Part A&B | Comparison of results between baseline and week 12.
  Cognitive functions are measured using digitized cognitive tests selected for depression in cooperation with Mindmore.
Cognitive function: Trail Making Test Part A&B | Comparison of results between baseline and year 1.
  Cognitive functions are measured using digitized cognitive tests selected for depression in cooperation with Mindmore.
Cognitive function: Symbol Digit Modalities Test | Comparison of results between baseline and week 12.
  Cognitive functions are measured using digitized cognitive tests selected for depression in cooperation with Mindmore.
Cognitive function: Symbol Digit Modalities Test | Comparison of results between baseline and year 1.
  Cognitive functions are measured using digitized cognitive tests selected for depression in cooperation with Mindmore.
Cognitive function: Corsi Block-Tapping Test forward | Comparison of results between baseline and week 12.
  Cognitive functions are measured using digitized cognitive tests selected for depression in cooperation with Mindmore.
Cognitive function: Corsi Block-Tapping Test forward | Comparison of results between baseline and year 1.
  Cognitive functions are measured using digitized cognitive tests selected for depression in cooperation with Mindmore.
Cognitive function: Rey Auditory Verbal Learning Test | Comparison of results between baseline and week 12.
  Cognitive functions are measured using digitized cognitive tests selected for depression in cooperation with Mindmore.
Cognitive function: Rey Auditory Verbal Learning Test | Comparison of results between baseline and year 1.
  Cognitive functions are measured using digitized cognitive tests selected for depression in cooperation with Mindmore.
Cognitive function: Stroop test | Comparison of results between baseline and week 12.
  Cognitive functions are measured using digitized cognitive tests selected for depression in cooperation with Mindmore.
Cognitive function: Stroop test | Comparison of results between baseline and year 1.
  Cognitive functions are measured using digitized cognitive tests selected for depression in cooperation with Mindmore.
Clinical Global Impression (CGI) severity scale | Up to 1 year from baseline.
  Clinician's impression of total severity of the mental illness. Scale between 0 and 7, higher point indicates worse outcome.
Posttraumatic Stress Disorder Checklist (PCL-5) | Up to 1 year from baseline.
  Measures symptoms in posttraumatic stress disorder. Total points 0-80, higher point indicates worse outcome.
Adult ADHD Self-Report Scale (ASRS) | Up to 1 year from baseline.
  Measures symptoms in attention deficiency and hyperactivity disorder (ADHD). Minimum 0 point to maximum 72 points. Higher point indicates worse outcome.
Perceived Stress Scale (PSS-14) | Up to 1 year from baseline.
  Measures perceived stress. Minimum 0 point to maximum 56 points. Higher point indicates worse outcome.
EuroQol-Health-Related Quality of Life (EQ-5D-5L) | Up to 1 year from baseline.
  Assesses the current overall health related to wellbeing and function experienced by the patient.
  The questionnaire consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  The EQ visual analogue scale (EQ VAS) records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine' between 0 and 100. The higher point indicates better outcome.

OTHER OUTCOMES:
Changes in gut microbiomes | Up to 1 year from baseline.
  The fecal samples will be analyzed for microbial composition using 16S microbiome analysis, metabolomics and Next Generation Sequencing.
Investigation of inflammatory biomarkers profile | Up to 1 year from baseline.
  Plasma and serum samples derived from the participants will be submitted for proteomics analyses to identify one or more plasma/serum proteins whose concentration over the course of the study varies in relation to the treatment response.
Investigation of fatty acid profiles | Up to 1 year from baseline.
  A fatty acid profile in the serum or plasma will be analyzed using gas chromatography coupled to mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Freund-Levi, MD, PhD, Principal Investigator — Region Örebro County/Örebro University
Locations (1):
- Department of Psychiatry, University hospital Örebro, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjorngrim S, van den Hurk W, Betancort M, Machado A, Lindau M. Comparing Traditional and Digitized Cognitive Tests Used in Standard Clinical Evaluation - A Study of the Digital Application Minnemera. Front Psychol. 2019 Oct 18;10:2327. doi: 10.3389/fpsyg.2019.02327. eCollection 2019. PMID 31681117